CLINICAL TRIAL: NCT06379165
Title: Efficacy and Safety Study of Meloxicam Nanocrystal Injection for the Treatment of Moderate to Severe Pain After Abdominal Surgery - a Multicenter, Randomized, Double-blind, Placebo-parallel Controlled, Phase III Clinical Trial
Brief Title: Efficacy and Safety Study of Meloxicam Nanocrystal Injection for the Treatment of Moderate to Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYH9015-002
Record Dates: First submitted 2023-01-28; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meloxicam Nanocrystal Injection (Experimental): The eligible subjects will receive Meloxicam Nanocrystal Injection, administered as 30 mg (1 mL) every 24 h for 2 doses.
  Interventions: Drug: Meloxicam Nanocrystal Injection
- Placebo (Placebo Comparator): The eligible subjects will receive Placebo, administered as 1 mL Placebo every 24 h for 2 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Meloxicam Nanocrystal Injection — 30 mg (1 mL), once daily, by intravenous infusion
  Arms: Meloxicam Nanocrystal Injection
Drug: Placebo — 1 mL Placebo, once daily, by intravenous infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of meloxicam nanocrystal injection in subjects with moderate to severe pain after abdominal surgery.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, placebo-controlled multicenter study will be conducted to evaluate the efficacy and safety of meloxicam nanocrystal injection in subjects with moderate to severe pain after abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ age ≤ 65 years, regardless of gender.
2. Elective abdominal surgery under general anesthesia.
3. ASA score of grade 1-3.
4. 18 kg/m^2 < BMI < 30 kg/m^2.
5. NRS score of ≥ 4 within 3 hours after the end of surgery (last suture).
6. Able to understand the study process and the use of pain scales, and able to communicate effectively with study personnel.
7. Written informed consent signed by subject or legal representative.

Exclusion Criteria:

1. Abnormal liver function: ALT and/or AST > 2 × ULN, or TBIL ≥ 2 × ULN.
2. Renal impairment (blood creatinine > 1.5 × ULN), or dialysis treatment within 28 days prior to the surgery.
3. Subjects at high risk of bleeding, including subjects with congenital bleeding disorders (e.g., hemophilia), thrombocytopenic subjects (platelet count less than 50 × 10^9/L), subjects with abnormal platelet function (e.g., idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital abnormal platelet function), or subjects with any clinically significant active bleeding.
4. Abnormal coagulation (PT>ULN+3s and/or APTT>ULN+10s).
5. Subjects with a history of severe gastrointestinal disease (e.g. ulcers, bleeding and perforation, etc.) within 1 year prior to randomization that may be worsened by the administration of NSAIDs-like drugs.
6. Myocardial infarction or coronary artery bypass grafting within 1 year prior to randomization.
7. Abnormal clinically significant 12-lead ECG during the screening period and judged by the investigator to be inappropriate for participation in this trial.
8. Combination of severe liver, kidney, cardiovascular, cerebrovascular, or metabolic system disease, which is judged by the investigator to be inappropriate for participation in this trial.
9. Subjects with combined neurological or psychiatric disorders such as migraine and seizures, which have been judged by the investigator to affect the evaluation of the efficacy of the trial drug.
10. Subjects with hypertension whose blood pressure is not satisfactorily controlled by antihypertensive medication (screening period sitting systolic blood pressure ≥ 160 mmHg, and/or screening period diastolic blood pressure ≥ 100 mmHg).
11. Sitting systolic blood pressure ≤ 90 mmHg at screening.
12. Subjects with diabetes mellitus whose blood glucose is not satisfactorily controlled (random blood glucose ≥ 11.1 mmol/L during the screening period).
13. Subjects with advanced malignancy or malignancy with extensive metastases.
14. Combined with other physical pain conditions that may confound postoperative pain evaluation.
15. Subjects with known hypersensitivity to meloxicam, any of the excipients in the study drug, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs), any perioperative drug use, or other history of anaphylactic reactions.
16. Subjects with alcohol or drug dependence within 3 months prior to screening and/or subjects whose alcohol, drug, or medication withdrawal may interfere with efficacy and safety evaluations during the study period.
17. Subjects who have undergone abdominal surgery within 6 months prior to randomization.
18. Subjects who have participated in other clinical trials and received the test drug/test device within 3 months prior to randomization.
19. Subjects with contraindications to investigational drugs, standard anesthetic practices.
20. Women who are pregnant or breastfeeding.
21. Other reasons that the investigator deems inappropriate for participation in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
PID24 (Time Weighted Sum of Pain Intensity Difference Over 24 Hours Post-Dose) | 24 hours after first dose
  The primary efficacy variable was the Pain Intensity (PI) measured by the Numerical Rating Scale (NRS); a scale from zero to 10 on which subjects circled a single number to indicate current pain level, with zero representing "No Pain" and 10 representing "Worst Possible Pain".

SECONDARY OUTCOMES:
TOTPAR (time-weighted sum of pain relief scores): TOTPAR12, TOTPAR18, TOTPAR24, TOTPAR48. | 0-48 hours after the first dose
  pain relief intensity was recorded using a Likert Scale (Range 0-4) where 0 equates to no pain relief (worse), and 4 equates to the completely pain relief intensity (better). pain relief intensity scores were to be recorded at the following time points: 0.25, 0.5, 1, 1.5, 2 ，3，4，6 ，8，10，12，14，16，18，24，30，36，42 and 48hours post Dose 1. pain relief intensity at each time point were calculated and a time weighted summed pain relief intensity (TOTPAR) was then calculated. Time weighted TOTPAR calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A bigger TOTPAR value was better.
SPID2、SPID6、SPID12、SPID18、SPID18-24、SPID24-48、SPID42-48、SPID48 | 0-48 hours after the first dose
  Pain intensity was recorded using a Numeric Pain Rating Scale (Range 0-10) where 0 equates to no pain (better), and 10 equates to the worst pain imaginable (worse). Pain intensity scores were to be recorded at the following time points: 0.25, 0.5, 1, 1.5, 2 ，3，4，6 ，8，10，12，14，16，18，24，30，36，42 and 48hours post Dose 1. Pain intensity differences from baseline at each time point were calculated and a time weighted summed pain intensity difference (SPID) was then calculated. Time weighted SPID calculations were computed by multiplying a weight factor to each score prior to summation. The weight factor at each time point was the time elapsed since the previous observation. A smaller SPID value (i.e. more negative) was better.
Time to the first dose of the remedial analgesia | 0-48 hours after the first dose
Number of times of remedial analgesia administered 0-24h and 24-48h after the first dose | 0-48 hours after the first dose
Proportion of subjects requiring remedial analgesia | 0-48 hours after the first dose
The total amount of remedial analgesia used 24 h and 48 h after the first dose | 0-48 hours after the first dose
The subject's analgesic treatment satisfaction score (0-4 point categorical scale score) | 48 hours after the first dose
  The subject's analgesic treatment satisfaction score was recorded using a Likert Scale (Range 0-4), A bigger value was better.
The investigator's satisfaction score (0-4 point categorical scale score) for the subject's analgesic treatment | 48 hours after the first dose
  The investigator's satisfaction score was recorded using a Likert Scale (Range 0-4), A bigger value was better.

CONTACTS AND LOCATIONS:
Overall Officials: Chen xiangdong, Principal Investigator — Union Hospital of Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, China

IPD SHARING:
Plan to Share IPD: No